CLINICAL TRIAL: NCT06964763
Title: Laser Ablation Versus Fibrin Glue in Mini-invasive Pilonidal Sinus Disease Surgery: a Prospective Randomized Controlled Trial
Brief Title: A Trial in Mini-invasive Pilonidal Sinus Disease Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Kethe Hermunen, Principal Investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS/2951/2021
Record Dates: First submitted 2025-04-23; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Pilonidal Disease
Keywords: pilonidal sinus disease; laser ablation; fibrine glue; randomized trial; prospective study
MeSH Terms: interventions — Laser Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group 1 (Active Comparator): surgery + laser ablation
  Interventions: Procedure: surgery + laser
- study group 2 (Active Comparator): surgery + fibrine glue
  Interventions: Procedure: surgery + fibrine glue

INTERVENTIONS:
Procedure: surgery + laser — laser
  Arms: study group 1
Procedure: surgery + fibrine glue — fibrine glue
  Arms: study group 2

SUMMARY:
Pilonidal sinus disease is a chronic acquired disease leading to significant morbidity and healthcare costs in young man and women. Despite different treatment methods, the disease relatively often leads to postoperative complications and recurrence.(8). Advantages of mini-invasive techniques include: quicker recovery and earlier return to work and high patient satisfaction. Randomized studies are rare and this applies especially to newer mini-invasive techniques. The purpose of the investigators prospective study is to randomly compare the mini-invasive laser ablation technique to the mini-invasive fibrin glue treatment in pilonidal sinus disease surgery.

DETAILED DESCRIPTION:
This is a multicenter study comparing two mini-invasive treatmnet options in pilonidal sinus disease. The study is carried out in four hospitals in Uusimaa county of Finland (Jorvi hospital, Porvoo hospital, Lohja hospital and Hyvinkää hospital). Patients, who are 18 or above, with a symptomatic primary pilonidal sinus disease are eligible for the study. On the day of surgery, the patient is randomly assigned to one of the two surgery groups. The main variable of our study is the healing rate at 2 months after surgery. Other variables to be studied are: postoperative complications, length of sick leave, time for returning to everyday life, recurrence rate and the effects of PSD and PSD surgery on the patient's quality of life. A cost analysis will be performed. Risk factors such as overweight, pubic hair, smoking and associated diseases such as diabetes will also be analyzed. According to the power calculation, the investigators need 94 patients in each group to ensure the success of the study.

ELIGIBILITY:
Inclusion Criteria:

* primary pilonidal sinus disease
* age 18 and above

Exclusion Criteria:

* recurrent pilonidal sinus disease
* age under 18
* inability to understand Finnish or Swedish (the questionnaires are in Finnish and Swedish only, the two official languages of Finland)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2029-06-17 (Estimated); Study Completion 2029-12-17 (Estimated)

PRIMARY OUTCOMES:
Healing rate | 2 months after surgery
  Healing rate will be assessed by a questionnaire and a phone call
Quality of life | 2 months after surgery
  Quality of life will be assessed by a questionnaire, the RAND 36-Item Health Survey

SECONDARY OUTCOMES:
Recurrence rate | 1, 3 and 5 years after surgery
  Follow-up at 1, 3 and 5 years by assessing electronic medical records to reveal recurrences
Cost analysis | At 2 months after surgery
  Compare the price for the two surgical treatments
Postoperative complications | 2 - 3 months after the surgery
  Postoperative complications will be assessed by a phone call and clinical examination
Sick leave | 2 months and 1 year after surgery
  Length of sick leave will be assessed by a questionnaire and medical records
Recovery time | 2 months and 1 year after surgery
  The time it has taken fot the patient to return to everyday life is assessed by a questionnaire and through medical records

CONTACTS AND LOCATIONS:
Overall Officials: Pauli Puolakkainen, Professor, Study Director — University of Helsinki, Department of Surgery
Locations (1):
- HUS Vatsakeskus Abdominal Center of Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided
We have not yet discussed this within the study group